CLINICAL TRIAL: NCT03055910
Title: A Fax-based Registry Regarding Clinical Indications, Complication Rates and Management Consequences of Invasive Fractional Flow Reserve Measurements
Brief Title: Fractional Flow Reserve Fax Registry
Acronym: F(FR)²
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: FFR_01_2017
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve Measurement — Wire-based invasive measurement of the fractional flow reserve in the context of coronary angiography and percutaneous coronary intervention in order to assess the hemodynamic relevance of coronary artery stenoses

SUMMARY:
The Fractional Flow Reserve Fax Registry is an investigator-initiated, real-world registry to analyze the use of fractional flow reserve (FFR) measurements in clinical practice in cardiac catheterization laboratories in Germany. The registry aims to collect the data of 2000 patients who underwent FFR recordings for clinical reasons. The main outcome parameter is the frequency of coronary revascularization following FFR. Secondary outcome parameters include the distribution of quantitative FFR results in clinical practice, the influence of intracoronary versus intravenous adenosine on the distribution of FFR results, the rate of complications as a result of FFR measurements, the average number of FFR wires needed per patient. Since the study will include a large number of patients who undergo i.c. administration of adenosine and a large number of patients who undergo i.v. administration of adenosine, it will be possible to analyze whether the route of adenosine administration is an independent predictor of the FFR result.

DETAILED DESCRIPTION:
Patient Inclusion Criteria

All patients who undergo measurement of the Fractional Flow Reserve using intracoronary pressure measurements for clinical reasons are eligible for inclusion.

There are no exclusion criteria.

Methods

Following a clinically indicated FFR measurement, patient data and data concerning angiographic stenosis severity as well as anatomic location of the interrogated lesion, method of adenosine administration, and FFR result are documented in a paper form. The form contains no patient data except age and gender as well as the cath lab identifying number and the serial number of the used FFR wire(s). The paper form is transmitted by fax to the central study site at Erlangen University where data will be stored and all evaluations will be performed.

Recruitment period

Recruitment starts March 1, 2017 and will be terminated after 2000 patients have been included.

Number of patients

2000 patients will be included.

Outcome parameters

The main outcome parameter is the frequency of coronary revascularization following FFR.

Secondary outcome parameters include the distribution of quantitative FFR results in clinical practice, the rate of complications as a result of FFR measurements, and the average number of FFR wires needed per patient, as well as the influence of i.c. versus i.v. administration of adenosine on the distribution of obtained FFR results.

All outcome parameters will be determined immediately after the end of invasive coronary angiography (and coronary intervention, if performed) in each patient (day 0). No follow-up will be performed.

Institutional Review Board (IRB)

The study protocol has been approved by the IRB of the Faculty of Medicine, University of Erlangen-Nürnberg (File Number 4_15B). Patient consent has been waived since data will be completely anonymized and no study-specific interventions are performed.

Primary Investigator

The study primary investigator is

Stephan Achenbach

Department of Cardiology

University of Erlangen

Ulmenweg 18

91054 Erlangen

Germany

The study co-primary investigator is

Helge Möllmann

Department of Cardiology

Johannes Hospital Dortmund

Johannesstraße 9-13

44137 Dortmund

Germany

Sponsor

The study is sponsored by the University Hospital Erlangen, Department of Cardiology. It is financed through a restricted grant by Abbott Vascular

ELIGIBILITY:
Inclusion Criteria:

* invasive fractional flow reserve measurement is performed for clinical reasons

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with known or suspected coronary artery disease in whom invasive fractional flow reserve measurement is performed for clinical reasons in the context of coronary angiography or percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Revascularization | 1 hour
  Rate of revascularization following measurement of the fractional flow reserve

SECONDARY OUTCOMES:
Complications | 1 hour
  Complication attributable to the invasive measurement of fractional flow reserve
Number of wires | 1 hour
  Number of FFR wires used per patient
Administration route | 1 hour
  Average FFR values obtained in the cohort when using intracoronary or intravenous injection of adenosine

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Achenbach, MD, Principal Investigator — Friedrich Alexander University Erlangen-Nuremberg
Locations (2):
- Germany (2):
  - St. Johannes Hospital, Dortmund
  - University Hospital, Erlangen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altstidl JM, Achenbach S, Feyrer J, Nazli JB, Marwan M, Gaede L, Mollmann H, Giesler T, Rittger H, Pauschinger M, Rudolph TK, Moshage W, Bruck M, Trobs M. Use of coronary physiology to guide revascularization in clinical practice: results of the F(FR)2 registry. Clin Res Cardiol. 2024 Jul;113(7):1081-1091. doi: 10.1007/s00392-024-02463-w. Epub 2024 Jun 4. PMID 38832995